CLINICAL TRIAL: NCT04683016
Title: Disease Perception and Oral Health Impact Profile (OHIP) Before and After Non-surgical Periodontal Treatment
Status: Completed | Type: Observational
Sponsor: University of Siena (Other)
Responsible Party: Principal Investigator, Nicola Discepoli, Professor, University of Siena
Other Study IDs: QU001
Record Dates: First submitted 2020-10-24; First posted 2020-12-24 (Actual); Last update posted 2020-12-24 (Actual); Status verified 2020-12

CONDITIONS: Periodontitis
Keywords: Oral Health Impact Profile 14; OHIP 14; non surgical periodontal treatment; brief-Illness Perception Questionnaire
MeSH Terms: conditions — Periodontitis | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Periodontitis patients: Patients with a diagnosis of periodontitis, irrespective of its stage and grade.
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — Patients will be asked two sets of questions:
  * questionnaire about their perception of periodontal disease (Brief Illness Perception Questionnaire; 9 questions, answers will be registered on a scale of 0 to 10);
  * Oral Health Impact Profile 14 (OHIP-14) questionnaire.
  All these two sets of questions will be asked before and after non surgical periodontal therapy

SUMMARY:
The presence of periodontal diseases in patients has been associated to a worsened quality of life overall. Many different indices have been proposed over time in order to evaluate patient's centred outcomes. In particular, the most thorough questionnaire proposed so far is the Oral Health Impact Profile 49 (OHIP-49), which is composed of 49 questions. Despite its validity being unquestionable, OHIP-49 was found to be too time-consuming for the clinical scenario and, therefore, its shortened 14-question version has been proposed. A more in-depth knowledge of how these parameters change before and after periodontal treatment could enable clinicians to tailor the treatment plan according to the patients' needs.

ELIGIBILITY:
Inclusion Criteria:

* patients being at least 18 years old
* Patients with a diagnosis of Periodontitis

Exclusion Criteria:

* diagnosis Gingivitis
* diagnosis of periodontal health
* inability or unwillingness to give informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with a diagnosis of Periodontitis will be eligible for the inclusion in the study.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Change in Brief Illness Perception Questionnaire (Brief IPQ) before and after non-surgical periodontal treatment | The questionnaire will be carried out at baseline and re-evaluation (3 months after non-surgical periodontal treatment). The change in the Brief IPQ values at baseline and after 3 months will be considered as the primary outcome measure.
  Brief Illness Perception Questionnaire consists of 9 questions, each one evaluated on a scale of 0 to 10 (minimum score of 0, maximum score of 90). Higher scores mean a higher patient's perception of the disease (higher scores mean worse outcome).
Change in Oral Health Impact Profile 14 before and after non-surgical periodontal treatment | The questionnaire will be carried out at baseline and re-evaluation (3 months after non-surgical periodontal treatment). The change in the OHIP-14 values at baseline and after 3 months will be considered as the primary outcome measure.
  14 questions about the impact of oral health on the quality of life; each question will be evaluated on a scale of 1 to 5 (minimum score of 0, maximum score of 70). Higher scores mean that patient's oral health impacts more significantly on their quality of life (higher scores, worse outcomes).

SECONDARY OUTCOMES:
Change in Full Mouth Bleeding Score (FMBS) before and after non-surgical periodontal treatment | FMBS will be calculated at baseline and re-evaluation (3 months after non-surgical periodontal treatment). The change in the FMBS at baseline and after 3 months will be considered as the secondary outcome measure.
  Full Mouth Bleeding Score will be calculated as the percentage of sites with Bleeding on Probing on the total number of sites (percentage ranging between 0% and 100%). Higher scores of FMBS mean more periodontal inflammation and therefore worse oral health (higher scores of FMBS, worse outcomes).

CONTACTS AND LOCATIONS:
Locations (1):
- AOUS, Siena, Italy